CLINICAL TRIAL: NCT05786534
Title: Therapeutic Potential of Green Seaweed, Ulva Lactuca, Against Metabolic Syndrome
Brief Title: Therapeutic Effect of Green Seaweed Against Metabloc Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Asif Ali, Researcher, University of Veterinary and Animal Sciences, Lahore - Pakistan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Green Seaweed
Record Dates: First submitted 2023-03-03; First posted 2023-03-27 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Hypertension; Diabetes; Obesity; Dyslipidemia; Seaweed
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Diabetes Mellitus; Obesity; Dyslipidemias

STUDY DESIGN:
Intervention Model Description: Case Control Study
Masking Description: Participants groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Metabolic Syndrome patients (Experimental): Green seaweed Ulva Lactuca is used for preventing symptoms in Metabolic Syndrome patients
  Interventions: Dietary Supplement: Green Seaweed

INTERVENTIONS:
Dietary Supplement: Green Seaweed — 400 mg per day
  Other Names: Ulva Lactuca

SUMMARY:
Metabolic syndrome is a major concern worldwide and in Pakistan as well. Metabolic syndrome is a pathologic condition which includes abdominal obesity, insulin resistance, hypertension and hyperlipidemia. Seafood consumption has been linked to reduced risk of many health conditions including altered blood profile. Green seaweed is known to have a potential in optimizing the blood profile and so, it is helpful in reducing the risk of metabolic syndrome by playing a role in preventing obesity, hyperglycemia, high blood pressure and altered lipid profile. Green seaweed (Ulva Lactuca) powder will prove to have therapeutic potential against obesity, hypertension, glucose intolerance and dyslipidemia.

DETAILED DESCRIPTION:
Metabolic syndrome is a major concern worldwide and in Pakistan as well. Metabolic syndrome is a pathologic condition which includes abdominal obesity, insulin resistance, hypertension and hyperlipidemia. Seafood consumption has been linked to reduced risk of many health conditions including altered blood profile. Green seaweed is known to have a potential in optimizing the blood profile and so, it is helpful in reducing the risk of metabolic syndrome by playing a role in preventing obesity, hyperglycemia, high blood pressure and altered lipid profile.

Statement of problem: The number of people with high LDL-cholesterol, body mass index and fasting plasma glucose levels has been increasing. These factors are promoting the risk of metabolic syndrome in Pakistan. 26-38% people in Pakistan are reported to be a patient of metabolic syndrome. Seaweed has shown to be protective against the syndrome in previous studies. The goal of this study is to check the role of green seaweed against metabolic syndrome.

Hypothesis: Green seaweed (Ulva Lactuca) has a potential to manage metabolic syndrome.

Objective: To assess the therapeutic effect of green seaweed (Ulva Lactuca) against metabolic syndrome.

Methodology: Green seaweed powder will be procured from Taokaenoi Food and Marketing Public Co., Ltd. (Thailand). The proximate analysis of the product will be performed and then capsules of powder will be prepared to be consumed by the participants. Total 40 subjects (20 in treatment group and 20 in control group) will be selected and green seaweed powder will be added in their diets (200mg twice a day). After a trial of 40 days, the patients will be assessed. Assessment will include anthropometric measurements, blood pressure, lipid profile analysis and total antioxidant capacity (TAC) which will be monitored before and after the trial and final,ly, the data collected will be analyzed by using SPSS 25 by paired sample t test. P value ≤ 0.05 will be considered significant.

Expected outcomes: Green seaweed (Ulva Lactuca) powder will prove to have therapeutic potential against obesity, hypertension, glucose intolerance and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25kg/m2
* Dyslipidemia
* Altered blood glucose level
* Age 30-55 ( male and female)

Exclusion Criteria:

* Thyroid disorder
* Liver disease
* Kidney disorder
* Cancer etc

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-09 (Actual); Primary Completion 2023-11-10 (Estimated); Study Completion 2023-11-10 (Estimated)

PRIMARY OUTCOMES:
Blood pressure will be assessed before and after the trial | 40 days
  The change in blood pressure, after consuming green seaweed powder for 40 days, will be assessed. The values will become close to optimized levels.
Lipid profile will be assessed before and after the trial | 40 days
  The improvement in lipid profile, after consuming green seaweed powder for 40 days, will be assessed. The values will become close to optimized values.
Fasting glucose level will be assessed before and after the trial | 40 days
  The change in fasting glucose levels will be assessed, after consuming green seaweed powder for 40 days. The values will become close to optimized levels.
Weight will be measured before and after the trial | 40 days
  The change in weight will be measured, after consuming green seaweed powder for 40 days. BMI will become close to normal range.

CONTACTS AND LOCATIONS:
Locations (1):
- Ashraf Hospital, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
All available data will be confidential

REFERENCES:
- [Result] Cardoso SM, Pereira OR, Seca AM, Pinto DC, Silva AM. Seaweeds as Preventive Agents for Cardiovascular Diseases: From Nutrients to Functional Foods. Mar Drugs. 2015 Nov 12;13(11):6838-65. doi: 10.3390/md13116838. PMID 26569268
- See also: Seaweeds as Preventive Agents for Cardiovascular Diseases — https://pubmed.ncbi.nlm.nih.gov/26569268/